CLINICAL TRIAL: NCT04654676
Title: The Effect of DPP4 Inhibitor on Glycemic Variability in Patients With Type 2 Diabetes Treated With Twice Daily Premixed Human Insulin
Brief Title: DPP4 Inhibitor on Glycemic Variability
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Malaysia Sarawak (Other)
Collaborators: Sarawak General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGH GV study
Record Dates: First submitted 2020-11-12; First posted 2020-12-04 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Vildagliptin — Vildagliptin added on to stable doses of pre-mixed insulin with or without metformin

SUMMARY:
The investigators conducted a prospective study in patients with T2DM on twice daily MHI with or without metformin therapy. Blinded continuous glucose monitoring was performed at baseline and following 6 weeks of Vildagliptin therapy.

DETAILED DESCRIPTION:
This was a prospective study involving adult patients with T2DM attending diabetes clinics in 2 state hospitals in Malaysia. Patients with HbA1c of 7-10% who were treated with stable dose of twice daily premixed human insulin (30% regular insulin, 70% Neutral Protamine Hagedorn) for at least 3 months, with or without metformin as combination therapy, were recruited. Consented participants attended a single education session with a diabetes nurse educator focusing mainly on self-monitoring of blood glucose (SMBG), hypoglycemia recognition and management, and the use of continuous glucose monitoring (CGM), before undergoing a 7 days blinded CGM (Medtronic MiniMed, Northridge, CA) to collect baseline GV data. The participants were instructed to perform SMBG 4 times daily for CGM calibration and record any symptomatic hypoglycemic episodes in the SMBG diary. Baseline demographic, insulin dosage as well as HbA1c and renal function were collected. The results of the CGM were blinded to the study participants and investigators till the end of the study.

Participants were then started on Vildagliptin (Novartis Pharma AG, Basel, Switzerland) for 6 weeks duration. The dose of Vildagliptin was determined based on calculated eGFR using MDRD (Modification of Diet in Renal Disease) IDMS (isotope dilution mass spectrometry) traceable formula. Vildagliptin 50 mg twice daily was prescribed for patients with eGFR ≥ 50 ml/min while patients with eGFR < 50 ml/min received Vildagliptin 50 mg daily as per prescription information recommendation. Drug accountability were assessed by tablet count. Throughout the study period, insulin doses were kept stable but may be adjusted by the investigators in the event of recurrent or severe hypoglycemia. The participants were also given the diabetes team's contact number for adjustment of insulin should they experience more frequent hypoglycemia with initiation of Vildagliptin, as per usual clinical practice.

A repeat 7 day CGM was performed after 6 weeks of Vildagliptin therapy. Changes in weight, insulin dosage and any symptomatic hypoglycemia episodes occurring during the study period were recorded. Data collected from the CGM device were analyzed with EasyGV software to derive the glycemic variability parameters. Primary outcome measures for GV were changes in mean amplitude of glycemic excursions (MAGE) and standard deviation of the mean glucose levels (SD). The investigators also examined other secondary GV measures including M value, mean absolute glucose (MAG), continuous overlapping net glycemic action (CONGA), low blood glucose index (LBGI), high blood glucose index (HBGI) and lability index (LI). In addition, quality of glycemic control with addition of DPP4-I treatment by assessing the % time in range (TIR) with blood glucose in target range of 3.9-10.0 mmol/L, % time above range (TAR), % time below range (TBR) and % of time spent in clinically significant level 2 hypoglycemia (blood glucose < 3.0 mmol/L regardless of symptoms) were explored. Area under the curve (AUC) above and below blood glucose target of 3.9 and 10.0 mmol/L respectively as well as glycemic estimate, i.e. estimated HbA1c (eA1c) from CGM data were also assessed before and after Vildagliptin treatment.

ELIGIBILITY:
Inclusion Criteria:

* HbA1c 7-10%
* Treated with stable dose of twice daily pre-mixed human insulin for at least 3 months, with or without metformin

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Changes in mean amplitude of glycemic excursions in mmol/L, Standard deviation of the mean glucose levels in mmol/L, M value in mmol/L, Mean absolute glucose in mmol/L, Continuous overlapping net glycemic action in mmol/L, Lability index in mmol/L | 12 months
  Glycemic variability

SECONDARY OUTCOMES:
Estimated HbA1c in %, % time in range (TIR) in %, % time above range (TAR) in %, % time below range (TBR) in %, % time below 3.0 mmol/L in % | 12 months
  Glycemic control
Low blood glucose index (LBGI) in mmol/L, High blood glucose index (HBGI) in mmol/L | 12 months
  Glycemic control
Area under curve above 10.0mmol/day, area under curve below 3.9mmol/day | 12 months
  Glycemic control

CONTACTS AND LOCATIONS:
Overall Officials: Florence Tan, Principal Investigator — Sarawak General Hospital
Locations (1):
- Sarawak General Hospital, Kuching, Malaysia

IPD SHARING:
Plan to Share IPD: No